CLINICAL TRIAL: NCT05595759
Title: The Effect of Creative Drama Training for Alcohol-Substance Addicted Male Patients on Attitudes Towards Violence Against Women: A Randomized Controlled Study
Brief Title: Violence Against Women in Patients With Alcohol Substance Addiction Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, HUMEYRA HANCER TOK, Head of Otolaryngology, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AİBÜ-HEM-HHT-01
Record Dates: First submitted 2022-09-27; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Woman Abuse; Addiction; Violence; Men
Keywords: Violence; Women; Addiction; Creative drama
MeSH Terms: conditions — Behavior, Addictive; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: In this study, the names of the patients hospitalized in the two wards will be sorted and numbered in alphabetical order. After the numbering process, the patients will be selected to the experimental and control group by using the "https://www.randomizer.org/" site by an independent specialist.
  In this study, the names of the patients hospitalized in the two wards will be sorted and numbered in alphabetical order. After the numbering process, the patients will be divided into an experimental and control group using the "https://www.randomizer.org/" site by an independent specialist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Male patients with a diagnosis of alcohol and substance abuse (Experimental): Male patients with a diagnosis of alcohol and substance abuse
  Interventions: Other: Violence against women education supported by creative drama
- Routine service operation (Other): Male patients with a diagnosis of alcohol and substance abuse
  Interventions: Other: Routine service operation

INTERVENTIONS:
Other: Violence against women education supported by creative drama — Violence against women supported by creative drama training will be applied to male patients diagnosed with addiction every day for 5 days.
  Arms: Male patients with a diagnosis of alcohol and substance abuse
Other: Routine service operation — No additional training will be applied to the control group and SAMBA trainings in the service operation will be applied.
  Arms: Routine service operation

SUMMARY:
This study was planned as a randomized controlled trial in order to determine the effect of creative drama training for alcohol-substance dependent male patients on their attitudes towards violence against women.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled trial in order to determine the effect of creative drama training for alcohol-substance dependent male patients on their attitudes towards violence against women.

The study was planned to be fully experimental. The participants to be included in the study will be selected from men who are followed up with a diagnosis of addiction in a mental health hospital. In the experimental group, male patients will be given violence against women training supported by creative drama five days a day. It will be used as an improved scale-measuring tool for women before and after the training. In the control group, the trainings applied in the service operation will be applied. It will be used as an improved scale-measuring tool for women before and after the training.

ELIGIBILITY:
Inclusion Criteria:

* Literate,
* Male inclusion,
* Have reached the age of 18,
* do not have an acute psychotic illness,
* Patients without symptoms of delirium tremens or intense withdrawal made up the study group of this study.

Exclusion Criteria:

* Illiterate,Woman,
* Have an acute psychotic illness,
* Delirium tremens or those with symptoms of intense withdrawal,
* Patients who did not agree to participate in the study were not included in this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Pretest final test scores on violence against women | 10 day
  Developed by Yalçın Kanbay in 2016, it is a 5-piece Likert type measurement tool consisting of two factors and 30 items. The scale has two sub-dimensions: "attitudes towards the body" and "attitudes towards identity". The total score of the scale is obtained by collecting the scores from two factors. On the scale, there are five answer options. In the scoring of the scale, each question is scored between 1-5. The high scores indicate that they are against violence against women, while the low scores indicate that they are not against violence against women. From the general scale, the lowest score is 30 and the highest score is 150. Kanbay found the Cronbach α value of the scale 0.86 for the overall scale. It is stated that the scale can be applied to individuals with at least primary school graduation and age between 15-65 years of age.
Pretest final test scores | 10 days
  Developed by Yalçın Kanbay in 2016, it is a 5-piece Likert type measurement tool consisting of two factors and 30 items. The scale has two sub-dimensions: "attitudes towards the body" and "attitudes towards identity". The total score of the scale is obtained by collecting the scores from two factors. On the scale, there are five answer options. In the scoring of the scale, each question is scored between 1-5. The high scores indicate that they are against violence against women, while the low scores indicate that they are not against violence against women. From the general scale, the lowest score is 30 and the highest score is 150. Kanbay found the Cronbach α value of the scale 0.86 for the overall scale. It is stated that the scale can be applied to individuals with at least primary school graduation and age between 15-65 years of age.

CONTACTS AND LOCATIONS:
Overall Officials: hümeyra Hançer tok, msc, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Mental Health and Diseases Hospital, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
WE WILL PREPARE THE STUDY AS A THESIS. THEN WE WILL TURN IT INTO A PUBLICATION IN AN INTERNATIONAL MAGAZINE
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: DATA WILL BE COLLECTED FOR 1 MONTH
Access Criteria: CAN BE CONTACTED THROUGH YÖK-THESIS CENTER

REFERENCES:
- [Background] ASAM. (2022, July 5). What is the definition of addiction? . File:///C:/Users/Lenovo/Desktop/B0209701-2099-441a-92c3-Eb60c4a387cb.Pdf.
- [Background] Bacchus LJ, Ranganathan M, Watts C, Devries K. Recent intimate partner violence against women and health: a systematic review and meta-analysis of cohort studies. BMJ Open. 2018 Jul 28;8(7):e019995. doi: 10.1136/bmjopen-2017-019995. PMID 30056376
- [Result] Aksoy, Y. D., Nacar, G., & Taşhan, S. T. (2018). Examine the attitudes toward spouse violence of health sciences faculty students Sağlık bilimleri fakültesi öğrencilerinin eş tarafından uygulanan şiddete ilişkin tutumları. Journal of Human Sciences, 15(2), 919-930
- [Derived] Tok HH, Kesgin MT. Effect of drama-education for alcohol/substance user on attitudes toward violence against women: randomized controlled design. BMC Public Health. 2025 May 15;25(1):1781. doi: 10.1186/s12889-025-23012-8. PMID 40375196

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT05595759/Prot_SAP_000.pdf
  • Informed Consent Form (2013-11-28): https://cdn.clinicaltrials.gov/large-docs/59/NCT05595759/ICF_001.pdf